CLINICAL TRIAL: NCT04378855
Title: Patient-Reported Outcomes in PHiladelphia-nEgative Cytogenetic mYeloproliferative Neoplasms (PROPHECY): A GIMEMA Observational Registry for Italian MPN Patients
Brief Title: Patient-Reported Outcomes in PHiladelphia-nEgative Cytogenetic mYeloproliferative Neoplasms (PROPHECY).
Acronym: PROPHECY
Status: Active, not recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: GIMEMA QoL-MPN 0118
Record Dates: First submitted 2020-04-28; First posted 2020-05-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Quality of life assessment

SUMMARY:
This study will ultimately aim at developing a GIMEMA platform for collecting HRQoL and symptom burden information on Italian patients with Philadelphia chromosome negative MPN. The main objective of the protocol is to improve our understanding of the impact of the disease and various treatments on patients-wellbeing, symptom burden and daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Polycythemia Vera (PV), Essential Thrombocythemia (ET) and Primary Myelofibrosis (pre-PMF, overt-PMF) and post-ET/post-PV Myelofibrosis (MF), (i.e. Philadelphia chromosome negative myeloproliferative neoplasm (MPN)) according to 2016 WHO classification.
* Known IPSS/IPSET/DIPSS risk score category at time of initial diagnosis of PV, ET and PMF, respectively.
* Initial diagnosis of MPN within one year before date of registration.
* Having a full baseline PRO Evaluation completed.
* Adult patients (≥ 18 years old).
* Written informed consent provided.

Exclusion Criteria:

* Having any kind of psychiatric disorder or major cognitive dysfunction problems hampering a self-reported evaluation.
* Not able to read and understand local language (i.e. Italian).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with myeloproliferative neoplasms (MPN)
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Compare HRQoL profiles of Philadelphia chromosome negative MPN patients with those of their peers in the general population | After 5 years from study entry
  To detect a baseline difference of at least 4 points between MPN patients and their peers in the general population in any of the following primary scales of the EORTC QLQ-C30 questionnaire: fatigue, global QoL/health status, physical, emotional and role functioning (all ranging from 0 to 100 points).

SECONDARY OUTCOMES:
Compare HRQoL profiles of Philadelphia chromosome negative MPN patients with those of their peers in the general population | After 5 years from study entry
  The same comparisons described for the primary endpoint will be performed on all other scales from EORTC QLQ-C30 questionnaire.
Compare HRQoL profiles of Philadelphia chromosome negative MPN patients with those of their peers in the general population | After 5 years from study entry
  The same comparisons described for the primary endpoint will be performed on all other scales from FACIT-Fatigue questionnaire.
MPN patients' baseline profiles of self-reported HRQoL | After 5 years from study entry
  To report MPN patients' baseline profiles of self-reported HRQoL and symptoms scores.
Prognostic value of baseline patients' self-reported fatigue | After 5 years from study entry
  To investigate the prognostic value of baseline patients' self-reported fatigue from EORTC QLQ-C30
Prognostic value of baseline patients' self-reported HRQoL | After 5 years from study entry
  To investigate the prognostic value of baseline patients' self-reported HRQoL
Relationship between pruritus and HRQoL. | After 5 years from study entry
  To investigate the relationship between Pruritus as assessed by MPN-SAF TSS questionnaire and HRQoL.
Patterns over time of HRQoL | After 5 years from study entry
  To estimate and compare patterns over time of HRQoL (outcome measures: EORTC QLQ-C30, FACIT-Fatigue, MPN-SAF TSS and FACIT-TS-G) of PT, EV and PMF patients.
Prognostic patient-based index | After 5 years from study entry
  To devise a prognostic patient-based index.
Physicians' and patients' preferences for involvement in treatment decision-making | After 5 years from study entry
  To assess physicians' and patients' preferences for involvement in treatment decision-making, as assessed by the CPS Questionnaire, across different risk groups and examine relationships between preferences for involvement and patient characteristics.
Relationship between self-reported satisfaction with care with other HRQoL outcomes. | After 5 years from study entry
  To investigate the relationship, in MPN patients, between self-reported satisfaction with care as assessed by the FACIT-TS-G questionnaire and its relationship with other HRQoL outcomes.

CONTACTS AND LOCATIONS:
Locations (25):
- Italy (25):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Asl Di Asti, Ospedali Riuniti - Presidio Ospedaliero Cardinal G. Massaia - Sc Oncologia, Asti
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Irccs Oncologico Istituto Tumori Giovanni Paolo Ii - Bari - Uo Ematologia, Bari
  - Istituto di Ematologia "Lorenzo e A. Seragnoli", Bologna
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - Azienda Ospedaliera "S.Gerardo", Monza
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - .C.D.U. Ematologia - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - C.R.O.B. - I.R.C.C.S. - Rionero in Volture - Uoc Ematologia, Rionero in Vulture
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Asl to 2, Torino Nord Emergenza San Giovanni Bosco - Ssd Ematologia, Torino
  - Ospedale Mauriziano Umberto I - Torino - Scdu Ematologia, Torino

IPD SHARING:
Plan to Share IPD: No